CLINICAL TRIAL: NCT05130021
Title: A Phase 2 Study to Evaluate the Safety and Efficacy of Max-40279-01 in Patients With Advanced Colorectal Cancer
Brief Title: A Clincal Study of Max-40279-01 in Patients With Advanced Colorectal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Maxinovel Pty., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MAX-40279-005
Record Dates: First submitted 2021-11-10; First posted 2021-11-22 (Actual); Last update posted 2021-12-06 (Actual); Status verified 2021-11

CONDITIONS: Metastatic Colorectal Cancer
Keywords: metastatic colorectal cancer; pretreated
MeSH Terms: conditions — Colorectal Neoplasms | interventions — regorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Part 1;50mg (Experimental)
  Interventions: Drug: MAX-40279-01
- Part 1;70mg (Experimental)
  Interventions: Drug: MAX-40279-01
- Part 2;MAX-40279-01 (Experimental)
  Interventions: Drug: MAX-40279-01
- Part 2;regorafenib (Experimental)
  Interventions: Drug: regorafenib

INTERVENTIONS:
Drug: MAX-40279-01 — MAX-40279-01 50mg/70mg
  Arms: Part 1;50mg; Part 1;70mg; Part 2;MAX-40279-01
Drug: regorafenib — regorafenib
  Arms: Part 2;regorafenib

SUMMARY:
This include two parts, part 1 is a dose optimizing study and part 2 is a randomized, controlled study.

DETAILED DESCRIPTION:
This study is a study of Max-40279-01 in patients with advanced colorectal cancer. This study include two Parts, the Part 1 will assess the safety and efficacy of the preset two dose level of Max-40279-01, and recommend a dose level of Max-40279-01 for stage 2. The part 2 is a randomized, controlled study ,and designed to compare the efficacy and safety of max-40279-01 to regorafenib or best support care(BSC) in pretreated advanced colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Males and/or females over age 18
2. Histologically and/or cytologically documented local advanced or metastatic colorectal adenocarcinoma.
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
4. Expected survival >3 months.
5. previously treated with standard, approved therapies, including two lines of chemotherapy (fluoropyrimidine,oxaliplatin and irinotecan based), a biological VEGF inhibitor, and, if RAS wild-type, an EGFR inhibitor. Patients with MSI-H/MMR-deficient tumors also must have received an immune checkpoint inhibitor, if available and approved. In addition, patients with BRAF mutant tumors must also have received a BRAF inhibitor, if available and approved.
6. Signed informed consent form.

Exclusion Criteria:

1. Known uncontrolled or symptomatic central nervous system metastatic disease.
2. Adverse events (with exception of alopecia, peripheral sensory neuropathy grade ≤ 2 and those listed in specific exclusion criteria) from any prior anticancer therapy of grade >1 (National Cancer Institute Common terminology Criteria [NCI CTCAE] v.3.0) at the time of randomization.
3. Inadequate organ or bone marrow function.
4. Medical history of difficulty swallowing, malabsorption or other chronic gastrointestinal disease, or conditions that may hamper compliance and/or absorption of the tested product.
5. Pregnant or breast-feeding woman.
6. Known allergies, hypersensitivity, or intolerance to Max-40279-01 the excipients of these treatments The above information was not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2022-01-31 (Estimated); Primary Completion 2022-05-30 (Estimated); Study Completion 2023-10-31 (Estimated)

PRIMARY OUTCOMES:
Disease control rate (DCR)[Part 1] | Through study Part 1 completion, an average of 6 months
progress free survival(PFS)[Part 2] | Through study Part 1 completion, an average of 6 months

SECONDARY OUTCOMES:
Tmax | Approximately 6 months
  Time to maximum plasma concentration
Cmax | Approximately 6 months
  Maximum plasma drug concentration
AUC | Approximately 6 months
  Area under the time-concentration curve
Objective response rate (ORR) | 6 months (anticipated)
overall survival (OS) | 24 months
Safety and tolerability assessed by incidence and severity of adverse events | 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- The Sixth Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No